CLINICAL TRIAL: NCT06730529
Title: The Value of 68Ga-FAPI PET/CT in Preoperative Evaluation of Thyroid Cancer with Lymph Node Metastases
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Hu Jiajia, Deputy director, Ruijin Hospital
Other Study IDs: RuijinH 2024-498
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Thyroid Cancer
Keywords: Thyroid Cancer; 68Ga-FAPI; PET/CT
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients diagnosis of thyroid cancer with lymph node metastases

SUMMARY:
This study aims to investigate the value of 68Ga-FAPI in the preoperative evaluation of thyroid cancer of different pathologic types.

DETAILED DESCRIPTION:
The investigators will number all participants, create a medical record file, and record their basic information (gender, age) as well as contact information and medical history information. All participants will undergo a 68Ga-FAPI PET/CT before surgery. The imaging response measurements will be compared with the histopathological results as gold standard.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological and clinical diagnosis of thyroid cancer with lymph node metastases.
2. Signed and dated informed consent form.
3. Commitment to comply with research procedures and co-operation in the implementation of the full research process.
4. Aged 16-80 years old.

Exclusion Criteria:

1. Patients with serious illnesses that researchers consider unsuitable for participation in this clinical study. Such as severe heart and lung failure, severe bone marrow suppression, severe liver and kidney dysfunction, etc.
2. Intestinal perforation, complete intestinal obstruction.
3. Pregnant women and women who may be pregnant, women who are breastfeeding.
4. Non-compliant person.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Inpatients and outpatients at Ruijin Hospital who meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-11-29 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical staging of thyroid cancer with lymph node metastasis | Within 1 week after enrollment
  The value of 68Ga-FAPI PET/CT in the evaluation of thyroid cancer with lymph node metastases in clinical staging

SECONDARY OUTCOMES:
Standardized uptake value(SUV) | Within 1 week after enrollment
  SUV of 68Ga-FAPI uptake on PET/CT images for tumor lesions
Disease free survival | 3 years
  Disease free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital affiliated to Shanghai Jiao Tong University of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No